CLINICAL TRIAL: NCT07368517
Title: Effect of Dry Needling in the Treatment of Patients With Mechanical Neck Pain
Brief Title: Dry Needling for Mechanical Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dry Needling
Record Dates: First submitted 2026-01-16; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2018-05

CONDITIONS: Mechanical Neck Pain; Neck Pain; Musculoskeletal Disorders; Cervical Spine Dysfunction
Keywords: Mechanical Neck Pain; Dry Needling; Myofascial Trigger Points; Cervical Spine; Cervical Range of Motion; Physical Therapy
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases | interventions — Dry Needling; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned into two parallel groups. Group A will receive dry needling with neck exercises, and Group B will receive TENS, ultrasound, and neck exercises.
  Both groups will receive treatment three times per week for four weeks.
Masking Description: This is an open-label study. Both participants and care providers are aware of the assigned interventions due to the physical nature of the treatments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry Needling with Exercise (Experimental): Participants in this group will receive dry needling to the upper trapezius and deltoid muscles under aseptic conditions. Needles will be inserted 5-10 mm deep and held for approximately 30 seconds, then discarded.
  This intervention will be combined with a neck exercise program including chin-in exercises (3 sets × 10 repetitions, 5-second holds) and a muscle energy technique (3 repetitions per side, holding 5-10 seconds).
  Sessions: three per week for four weeks.
  Interventions: Other: Dry Needling with Exercise
- Conventional Physiotherapy with Exercise (Active Comparator): Participants in this group will receive conventional physiotherapy including transcutaneous electrical nerve stimulation (TENS) at 80-100 Hz, 100 µs pulse duration for 20 minutes, and pulsed ultrasound at 1 MHz, 1.0-1.5 W/cm² for 5 minutes.
  The same exercise program will be applied (chin-in and muscle-energy technique).
  Sessions: three per week for four weeks.
  Interventions: Other: Conventional Physiotherapy with Exercise

INTERVENTIONS:
Other: Dry Needling with Exercise — Manual therapy procedure using sterile, single-use needles inserted into the upper trapezius and deltoid muscles for approximately 30 seconds to reduce trigger point activity. Combined with neck exercises (chin-in and muscle-energy technique).
  Administered three times per week for four weeks.
  Arms: Dry Needling with Exercise
Other: Conventional Physiotherapy with Exercise — Standard physiotherapy treatment consisting of TENS (80-100 Hz, 100 µs, 20 min) and ultrasound (1 MHz, 1.0-1.5 W/cm², 5 min) combined with neck exercises (chin-in and muscle-energy technique).
  Administered three times per week for four weeks.
  Arms: Conventional Physiotherapy with Exercise

SUMMARY:
Mechanical neck pain is one of the most common musculoskeletal disorders among adults. It is characterized by pain and stiffness in the cervical region, often related to poor posture, repetitive movements, or prolonged sitting. The condition can lead to functional limitations and decreased quality of life.

This randomized controlled clinical trial aims to evaluate the effectiveness of dry needling therapy on pain intensity, cervical range of motion, and functional ability in patients with mechanical neck pain. Forty participants aged 25 - 65 years will be randomly assigned to two groups. Group A will receive dry needling combined with neck exercises, while Group B will receive transcutaneous electrical nerve stimulation (TENS), ultrasound, and the same neck exercise program. Both groups will undergo treatment three times per week for four weeks.

Primary outcomes include changes in the Neck Disability Index (NDI), pressure pain threshold (PPT) measured by algometer, and cervical range of motion (CROM). The study will determine whether dry needling provides superior clinical improvement compared with conventional electrotherapy and exercise.

DETAILED DESCRIPTION:
Mechanical neck pain (MNP) affects a large proportion of adults between 25 and 65 years of age. It is commonly associated with sustained poor posture, repetitive movement, or prolonged sitting, leading to muscular tightness and joint stiffness in the cervical region. Patients typically present with pain, limited cervical mobility, and decreased ability to perform daily activities.

Dry needling is a minimally invasive technique that involves inserting fine monofilament needles into myofascial trigger points to reduce muscle tension, improve circulation, and alleviate pain. It is increasingly used in physiotherapy practice as a targeted intervention for musculoskeletal pain conditions. By releasing taut muscle bands, dry needling is believed to normalize muscle tone and restore normal movement patterns.

The current randomized controlled trial is designed to assess the effectiveness of dry needling combined with therapeutic exercise compared with conventional physiotherapy including TENS, ultrasound, and the same exercise regimen. Forty participants with mechanical neck pain will be randomly allocated into two equal groups (n = 20 per group).

Group A (Experimental): Dry needling will be applied to the upper trapezius and deltoid muscles under aseptic technique. Each needle will be inserted 5 - 10 mm deep and retained for approximately 30 seconds. This intervention will be combined with a neck exercise program consisting of chin-in exercises (3 sets × 10 repetitions, 5-second hold) and a muscle-energy technique for the upper trapezius (3 repetitions per side, 5 - 10 second holds).

Group B (Active Comparator): Participants will receive TENS at 80 - 100 Hz frequency, 100 µs pulse duration for 20 minutes, and pulsed ultrasound at 1 MHz, 1.0 - 1.5 W/cm² for 5 minutes. The same chin-in and muscle-energy exercise protocol will be applied.

Both groups will receive three sessions per week for four weeks. Assessments will include:

Pain and disability using the Neck Disability Index (NDI).

Pressure pain threshold (PPT) using a handheld algometer.

Cervical range of motion (CROM) using a cervical range-of-motion device.

Outcomes will be recorded at baseline and after four weeks of treatment. It is hypothesized that dry needling will produce greater reductions in pain and disability and larger improvements in cervical motion compared with conventional therapy.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable individuals who provide written informed consent to participate in the study.
* Age between 25 and 65 years.
* Both male and female participants.
* Patients diagnosed with mechanical neck pain lasting more than three months.
* Presence of myofascial trigger points in the upper trapezius or cervical muscles confirmed by palpation.
* Ability to follow treatment instructions and attend all scheduled sessions.

Exclusion Criteria:

* History of neck surgery or cervical spine fracture.
* Previous dry needling or invasive therapy for neck pain in the past six months.
* History of neurological disorders (e.g., cervical radiculopathy, myelopathy).
* Current acute infection, skin disease, or open wound in the neck or shoulder region.
* Use of anticoagulant medication or any bleeding disorder.
* Pregnancy or suspected pregnancy.
* Any systemic illness (e.g., diabetes mellitus, rheumatoid arthritis) that may affect healing or pain perception.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-10-05 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Neck Disability Index (NDI) | Baseline and after 4 weeks of treatment
  The Neck Disability Index (NDI) is a 10-item self-reported questionnaire used to assess how mechanical neck pain affects daily activities. Each item is scored from 0 to 5, and total scores are converted to a percentage, with higher values indicating greater disability. It is a valid and reliable tool for monitoring functional improvement after physiotherapy interventions.
Change in Pressure Pain Threshold (PPT) | Baseline and after 4 weeks of treatment
  Pressure Pain Threshold (PPT) will be measured using a digital algometer. It represents the minimum pressure that elicits pain and provides an objective assessment of muscle tenderness and trigger point sensitivity. Higher values indicate reduced pain sensitivity. Measurements will be taken over the upper trapezius muscle in kg/cm².
Change in Cervical Range of Motion (CROM) | Baseline and after 4 weeks of treatment
  Cervical Range of Motion (CROM) will be assessed using a CROM device that quantifies cervical flexion, extension, lateral flexion, and rotation. Measurements will be taken in degrees. The device provides objective and reproducible data on cervical spine mobility and is used to evaluate the effect of treatment on movement limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of physical therapy, Deraya University, Minya, Menia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ebadi, S., Ansari, N. N., Naghdi, S., & Jalaie, S. (2018). The effect of therapeutic ultrasound on neck pain: A systematic review. Ultrasound in Medicine & Biology, 44(3), 566-576. https://doi.org/10.1016/j.ultrasmedbio.2017.11.014
- [Background] Audette, I., Dumas, J. P., Côté, J. N., & De Serres, S. J. (2019). Validity and between-day reliability of cervical range of motion measurements. Journal of Orthopaedic & Sports Physical Therapy, 49(7), 510-517. https://doi.org/10.2519/jospt.2019.8583
- [Background] Tousignant-Laflamme, Y., Boutin, A., Dion, A. M., & Vallée, C. A. (2017). Reliability and criterion validity of two applications of the cervical range of motion device. Physiotherapy Theory and Practice, 33(2), 140-150. https://doi.org/10.1080/09593985.2016.1271845
- [Background] Vaegter HB, Handberg G, Graven-Nielsen T. Similarities between exercise-induced hypoalgesia and conditioned pain modulation in humans. Pain. 2014 Jan;155(1):158-167. doi: 10.1016/j.pain.2013.09.023. Epub 2013 Sep 26. PMID 24076045
- [Background] Walton DM, Macdermid JC, Nielson W, Teasell RW, Chiasson M, Brown L. Reliability, standard error, and minimum detectable change of clinical pressure pain threshold testing in people with and without acute neck pain. J Orthop Sports Phys Ther. 2011 Sep;41(9):644-50. doi: 10.2519/jospt.2011.3666. Epub 2011 Sep 1. PMID 21885906
- [Background] Vernon H. The Neck Disability Index: state-of-the-art, 1991-2008. J Manipulative Physiol Ther. 2008 Sep;31(7):491-502. doi: 10.1016/j.jmpt.2008.08.006. PMID 18803999
- [Background] Navarro-Santana MJ, Sanchez-Infante J, Fernandez-de-Las-Penas C, Cleland JA, Martin-Casas P, Plaza-Manzano G. Effectiveness of Dry Needling for Myofascial Trigger Points Associated with Neck Pain Symptoms: An Updated Systematic Review and Meta-Analysis. J Clin Med. 2020 Oct 14;9(10):3300. doi: 10.3390/jcm9103300. PMID 33066556
- [Background] Liu L, Huang QM, Liu QG, Ye G, Bo CZ, Chen MJ, Li P. Effectiveness of dry needling for myofascial trigger points associated with neck and shoulder pain: a systematic review and meta-analysis. Arch Phys Med Rehabil. 2015 May;96(5):944-55. doi: 10.1016/j.apmr.2014.12.015. Epub 2015 Jan 7. PMID 25576642
- [Background] Gross AR, Paquin JP, Dupont G, Blanchette S, Lalonde P, Cristie T, Graham N, Kay TM, Burnie SJ, Gelley G, Goldsmith CH, Forget M, Santaguida PL, Yee AJ, Radisic GG, Hoving JL, Bronfort G; Cervical Overview Group. Exercises for mechanical neck disorders: A Cochrane review update. Man Ther. 2016 Aug;24:25-45. doi: 10.1016/j.math.2016.04.005. Epub 2016 Apr 20. PMID 27317503
- [Background] Blanpied PR, Gross AR, Elliott JM, Devaney LL, Clewley D, Walton DM, Sparks C, Robertson EK. Neck Pain: Revision 2017. J Orthop Sports Phys Ther. 2017 Jul;47(7):A1-A83. doi: 10.2519/jospt.2017.0302. PMID 28666405
- [Background] Cote P, Wong JJ, Sutton D, Shearer HM, Mior S, Randhawa K, Ameis A, Carroll LJ, Nordin M, Yu H, Lindsay GM, Southerst D, Varatharajan S, Jacobs C, Stupar M, Taylor-Vaisey A, van der Velde G, Gross DP, Brison RJ, Paulden M, Ammendolia C, David Cassidy J, Loisel P, Marshall S, Bohay RN, Stapleton J, Lacerte M, Krahn M, Salhany R. Management of neck pain and associated disorders: A clinical practice guideline from the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Eur Spine J. 2016 Jul;25(7):2000-22. doi: 10.1007/s00586-016-4467-7. Epub 2016 Mar 16. PMID 26984876